CLINICAL TRIAL: NCT01202851
Title: Biobehavioral Effects of Relaxation for Women With Breast Cancer Undergoing Radiotherapy
Brief Title: Relaxation for Women With Breast Cancer Undergoing Radiotherapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-0976; NCI-2012-01895 (Registry Identifier: NCI CTRP); 2T32CA009666-21 (NIH)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: radiotherapy; radiation therapy; stretching; relaxation; quality of life; QOL; fatigue; sleep disturbances; mental health; cost-effectiveness analysis; work productivity; home productivity; cortisol rhythmicity
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Parasomnias; Psychological Well-Being | interventions — Relaxation Therapy; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxation Group 1 (Experimental): Simple stretching exercises, specific breathing skills, and guided relaxation for 3 sessions, 3 times a week for 6 weeks. Each session should last about 60 minutes. Multiple questionnaires taken before, during and after radiotherapy/exercise intervention programs during course of study. 4 saliva samples per day for cortisol testing for 3 days before radiation therapy begins, for 3 days in the last week of radiation therapy, for 3 days in a row 3 months after radiation therapy ended, for 3 days in a row, for 6 months after radiation therapy ended, and for 12 months after radiation therapy ended.
  Interventions: Other: Relaxation Program; Behavioral: Questionnaires; Other: Saliva Testing
- Relaxation Group 2 (Experimental): Simple stretching exercises, specific breathing skills, and guided relaxation for 3 sessions, 3 times a week for 6 weeks. Each session should last about 60 minutes. Multiple questionnaires taken before, during and after radiotherapy/exercise intervention programs during course of study. 4 saliva samples per day for cortisol testing for 3 days before radiation therapy begins, for 3 days in the last week of radiation therapy, for 3 days in a row 3 months after radiation therapy ended, for 3 days in a row, for 6 months after radiation therapy ended, and for 12 months after radiation therapy ended.
  Interventions: Other: Relaxation Program; Behavioral: Questionnaires; Other: Saliva Testing
- Waitlist Control Group (WLC) (Other): Participants in this group given the option to take part in one of the two forms of relaxation (off study) after they finish their last questionnaire packet. 4 saliva samples per day for cortisol testing for 3 days before radiation therapy begins, for 3 days in the last week of radiation therapy, for 3 days in a row 3 months after radiation therapy ended, for 3 days in a row, for 6 months after radiation therapy ended, and for 12 months after radiation therapy ended.
  Interventions: Behavioral: Questionnaires; Other: Saliva Testing

INTERVENTIONS:
Other: Relaxation Program — 3 times a week, 60 minute sessions for 6 weeks.
  Arms: Relaxation Group 1; Relaxation Group 2
Behavioral: Questionnaires — Multiple questionnaires taken before, during and after radiotherapy/exercise intervention programs during course of study.
  Other Names: survey
Other: Saliva Testing — 4 saliva samples per day for cortisol testing for 3 days before radiation therapy begins, for 3 days in the last week of radiation therapy, for 3 days in a row 3 months after radiation therapy ended, for 3 days in a row, for 6 months after radiation therapy ended, and for 12 months after radiation therapy ended.

SUMMARY:
The goal of this behavioral research study is to compare two different forms of relaxation programs that will include stretching and relaxation techniques, in order to learn if and how well they may help to improve physical and emotional well-being. This will be tested in patients with breast cancer who are receiving radiation therapy. For comparison purposes, there will also be a group of participants that does not take part in the relaxation programs.

This is an investigational study. The relaxation programs are being compared for research purposes only.

An "assessment" is any time you complete a set of scheduled activities for this study, such as tests and questionnaires.

Up to 700 patients will take part in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
During the first visit, you will fill out questionnaires that ask about your sleeping habits, how you have been feeling, and the general quality of your life. This should take about 60-80 minutes.

Every day for the next 7 days, you will fill out a diary about your sleep. You will also wear an "actigraph" wrist watch 24 hours a day for these 7 days. The watch will collect data about your physical activity and sleeping habits.

You will also have an electrocardiogram (ECG - a test to measure the electrical activity of your heart) which will last about 10 minutes.

Study Groups:

After your first visit, you will be randomly assigned (as in the roll of dice) to 1 of 3 groups:

* Group 1 will take part in one type of relaxation program.
* Group 2 will take part in another type of relaxation program.
* Group 3 will not take part in either program but will complete some of the follow-up procedures. Participants in this group will be given the option to take part in one of the two forms of relaxation (off study) after they finish their last questionnaire packet.

You will have about a 1 out of 3 chance of being assigned to each group. The groups are randomly assigned, but it is also based on other factors such as your age and the status of the disease.

Sessions:

Groups 1 and 2:

You will take part in 3 sessions each week for the 6 weeks of radiation therapy, or 4-5 sessions each week for 4 weeks if your radiation therapy lasts only 4 weeks. You can choose any weekday (Monday through Friday). Each session should last about 60 minutes.

The sessions will be taught by an experienced, trained instructor, usually in groups of 2-5 participants. The movements are designed to be easy to follow. You will be able to work at your own pace.

Each session will be audio and video recorded. This is so the researchers can keep track of the quality of the sessions. The audio and video files are digital and will be deleted after all the data are studied.

Women in Groups 1 and 2 will be randomized to a maintenance intervention arm or a usual contact arm after the end of radiotherapy. If you are randomized to the maintenance intervention arm you will receive telephone counseling once a month after the end of your radiotherapy. You will also receive booster sessions once every 3 months post-radiotherapy, or at least when you come for your follow-up appointments.

Groups 1 and 2:

During the sessions, you will do simple stretching exercises, specific breathing skills, and guided relaxation. You will be asked to try and practice once a day for 12 months. You will be provided a DVD and an audio CD to help with your practice when you are not at the hospital.

Questionnaires and Study Procedures:

Groups 1 and 2:

Before your first session of the week except for week 1, Groups 1 and 2 will fill out a questionnaire about the relaxation program. This should take about 1-2 minutes.

During the middle of your radiation treatment period, you will have an ECG recorded before and after your classes. Each ECG will last about 10 minutes.

All Groups:

During the middle of your radiation treatment period, you will fill out a questionnaire that asks about any symptoms you may be having. This should take about 15 minutes. You will also have an ECG.

During your last week of radiation therapy, and at 3, 6, and 12 months after your radiation therapy ends, you will fill out a set of questionnaires. The questionnaires will be mostly the same as at your first study visit. This should take about 60-80 minutes. You will also have an ECG at these times.

Questionnaire packets will be mailed to your home by the research staff. After completing the questionnaires, you will return the completed questionnaire packet to the research staff via a pre-paid mailing envelope.

Every day for 7 days in a row, after every time you fill out the questionnaires, you will fill out another sleep diary. During these 7-day periods, you will wear an actigraph watch 24 hours a day to collect the same data as before. Each time, you will mail the actigraph watch back to MD Anderson in postage-paid envelopes that will be provided to you.

If your questionnaire responses show that you may be having emotional difficulties or depression, you will be provided with names of mental health providers in case you would like to receive mental health screening.

All participants will be asked not to do any other stretching/relaxation practices during the study.

Saliva Testing:

You will provide 4 saliva samples per day for cortisol testing on the following schedule:

* for 3 days before radiation therapy begins
* for 3 days in the last week of radiation therapy
* for 3 days in a row, 3 months after radiation therapy ended
* for 3 days in a row, 6 months after radiation therapy ended
* for 3 days in a row, 12 months after radiation therapy ended

To provide a saliva sample, you will chew on a cotton ball for a few seconds and then put the cotton in a small plastic tube. You will then mail the samples back to MD Anderson in postage-paid envelopes that will be provided to you. The tubes will also be provided at no cost to you. These saliva samples will be destroyed after being studied.

Length of Participation:

Your study participation will be over after you fill out the questionnaires 12 months after radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women with stage 0 - III breast cancer who will be undergoing daily adjuvant radiation for 4-6 weeks (patients only).
2. 18 years of age or older (patient and spouse/partner).
3. Able to read, write, and speak English or Spanish (patient and spouse/partner).

Exclusion Criteria:

1. Patients who have any major psychiatric diagnoses (e.g., schizophrenia, bipolar disorder).
2. Patients who have not undergone any surgical treatment for their cancer.
3. Patients with extreme mobility issues (e.g., unable to get in and out of a chair unassisted).
4. Patients who have practiced yoga or taken yoga classes in the year prior to study enrollment or who are currently engaged in a regular mind-body practice.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2011-02-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Relaxation Program | Prior to and during radiotherapy, through 6 week relaxation program and 12 months post radiotherapy
  Effectiveness of 6-week relaxation intervention evaluated by physical component scale scores during and after treatment, defined as Medical Outcomes Study 36-item short-form survey (SF-36).

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org